CLINICAL TRIAL: NCT02053311
Title: Orteronel Maintenance Therapy in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC) Previously Treated With Novel Hormonal Agents and Non-progressive Disease After Treatment With a Taxane: A Multicentre Randomized Double-blind Placebo-controlled Phase III Trial
Brief Title: Orteronel Maintenance Therapy in Patients With mCRPC Previously Treated With Novel Hormonal Agents
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to former trials, drug has not demonstrated a clinical profile sufficient to move forward in mCRPC
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAKK 08/13; 2013-004912-23 (EudraCT Number)
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; metastatic castration-resistant prostate cancer; maintenance therapy; orteronel; TAK-700
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Orteronel (Active Comparator): 300mg orteronel twice daily and best supportive care until disease progression
  Interventions: Drug: Orteronel
- Arm B: Placebo (Active Comparator): Placebo twice daily and best supportive care until disease progression
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orteronel — 300mg orteronel
  Other Names: TAK-700
  Arms: Arm A: Orteronel
Drug: Placebo — Placebo
  Arms: Arm B: Placebo

SUMMARY:
The main object of this multicenter, randomized, double-blind, placebo-controlled phase III trial is to assess impact of maintenance of orteronel on disease progression and hence on quality of life of patients with metastatic castration resistant prostate cancer pretreated with novel hormonal agents who have non-progressive disease after chemotherapy with a taxane.

DETAILED DESCRIPTION:
Background

One in six men will be diagnosed with cancer of the prostate during his lifetime. Accordingly, prostate cancer is the most common cancer amongst men in the western world. In Switzerland approx. 5'400 men are diagnosed with the disease and 1'300 die of prostate cancer every year. Prostate cancer represents 30% of all cancer diagnoses in men. Despite earlier detection and new treatments the life time risk to die of prostate cancer has remained stable at 3% since 1980.

In metastatic castration-resistant prostate cancer (with progression on antihormonal therapy) the primary standard therapy for a long time consisted of chemotherapy with docetaxel. It was recently shown that treatment with the novel androgen synthesis blocker, abiraterone (Zytiga) before chemotherapy can prolong survival. Abiraterone belongs to a group of agents that very effectively inhibits the androgen synthesis via blockade of the key enzyme cytochrome P-450c17 (CYP17).Similar results have been reported for the new androgen antagonist enzalutamide (Xtandi). Today, therefore, many patients with metastatic castration-resistant prostate cancer (mCRPC) first receive therapy with abiraterone or enzalutamide. After this, chemotherapy with docetaxel (Taxotere) or cabazitaxel (Jevtana) is usually administered if there is any further progression of the disease. After the end of chemotherapy, the patient is regularly checked and, in the event of disease progression, further treatments may be given. These could consist of renewed hormonal therapy or chemotherapy with cabazitaxel. Besides abiraterone, the medicine orteronel also acts by blocking testosterone production via the key enzyme CYP17. By selectively inhibiting the extragonadal synthesis of androgens in either the adrenal cortex or in prostate tumor cells, orteronel, a selective non-steroidal CYP17 inhibitor, may represent a new therapeutic option for patients with CRPC. Initial results have shown that orteronel effectively inhibits testosterone synthesis.

Hypothesis and aim of the study

Since various new options are available for treatment of castration-resistant prostate cancer at present, this raises the question as to the order in which these treatments should best be given. Initial results show that cross-resistance could develop between the new kinds of hormone therapy abiraterone and enzalutamide. There is evidence to suggest that any resistance to hormone treatments could be reversible as a result of prior treatment with chemotherapy. This study is designed to investigate this approach. It is also intended to investigate whether early use of the well-tolerated testosterone synthesis blocker orteronel in patients with mCRPC leads to an increase in the time to the progression of disease. Trials examining other advanced malignant diseases such as lung cancer have shown that initiating an effective treatment earlier in the disease course at the end of a first-line chemotherapy (so called switch maintenance therapy) is beneficial in terms of progression free survival (PFS) but also overall survival (OS). This may also hold true for early administration of antihormonal agents in patients with mCRPC.

Patients who have already received a novel hormonal therapy followed by chemotherapy with a taxane and have experienced a stabilization of disease on this regimen are included in the study. It is also intended to test whether this treatment has a positive influence on the quality of life of patients.

The aim of this trial is to test the hypothesis that using orteronel treatment immediately after cessation of chemotherapy with a taxane can prolong event-free survival (EFS), consequently maintains a good quality of life (QL) and could eventually also improve overall survival for the group of patients pretreated with novel hormonal agents.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Male patient 18 years or older
* WHO performance status of ≤2
* Adenocarcinoma of the prostate, histologically or cytologically confirmed
* Castration resistance: tumor progression after orchiectomy or during treatment with GnRH analogues (agonists or antagonists)
* Metastatic disease, radiographically documented (CT/MRI, bone scan)
* Total testosterone ≤ 50 ng/dL (≤ 1.7 nmol/L)
* Treatment with a CYP17 inhibitor or a novel antiandrogen (such as enzalutamide, ODM-201, ARN-509, but not restricted to) or the combination of both agents) for at least 8 weeks prior to one line of a taxane based chemotherapy.
* No evidence of disease progression after chemotherapy with docetaxel (cumulative dose of ≥ 450 mg/m2 or total dose ≥900mg) or cabazitaxel (cumulative dose of ≥150 mg/m2 or total dose ≥300mg)
* Non-surgically castrated patient agrees on ongoing use of GnRH analogues (agonists or antagonists) during the trial
* Laboratory values as specified below

  * Potassium ≥ 3.5 mmol/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L and platelet count ≥ 100 x 109/L
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Total bilirubin ≤ 1.5 x ULN (except for patient with Gilbert's disease ≤ 5.0 x ULN)
  * Estimated creatinine clearance using the Cockcroft-Gault formula > 40 mL/minute
* Planned start of trial treatment 2 to 8 weeks after last taxane dose
* Calculated ejection fraction of ≥ 50% or normal according to local standard by echocardiogram or by multiple gated acquisition (MUGA) scan.
* Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before expected start of treatment
* Patient is able and willing to complete Baseline QL questionnaire completed
* Patient is able and willing to swallow study drug as whole tablet
* Patient compliance and geographic proximity allow proper staging and follow-up
* Patient, even if surgically sterilized (i.e., status post vasectomy)

  * agrees to practice effective barrier contraception during the entire study treatment period and for 4 months after the last dose of study drug, or
  * agrees to practice true abstinence, when this is in line with the preferred and usual lifestyle of the patient.

Exclusion Criteria:

* Prior therapy with aminoglutethimide and/or ketoconazole
* Prior chemotherapy for prostate cancer within 12 months before enrollment except from chemotherapy with a taxane
* Retreatment with a taxane for metastatic prostate cancer after interruption of > 8 weeks
* Concurrent disease requiring higher doses of corticosteroid than the equivalent of 10 mg prednisone per day
* Known allergy and/or hypersensitivity and/or any known grade 4 toxicity to modern CYP17 inhibitors and to any of their components and GnRH
* Concurrent treatment with other experimental drugs or treatment in a clinical trial within 30 days prior to trial entry
* Presence of a small cell component in histological specimen
* Radiotherapy within the last 2 weeks before expected start of the trial treatment
* Known history of central nervous system (CNS) or spinal cord metastases
* Current spinal cord compression
* Diagnosis of or treatment for another systemic malignancy within 2 years before registration or patient previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any time are not excluded if they have undergone complete resection.
* History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade ≥ 3 (NCI CTCAE version 4.0) or thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events) or any other cardiac condition (e.g. pericardial effusion, restrictive cardiomyopathy) within 6 months before the first dose of study drug. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed
* New York Heart Association Class III or IV heart failure
* ECG abnormalities of:

  * Q-wave infarction, unless identified ≥ 6 months prior to registration
  * QTc interval > 460 msec
* Uncontrolled hypertension despite appropriate medical therapy (systolic blood pressure > 160 mm Hg or diastolic blood pressure > 90 mmHg) at 2 separate measurements no more than 60 minutes apart during the Screening visit).
* Likely inability (e.g. due to a Psychiatric disorder) to understand information on trial related topics, to give informed consent, to comply with the protocol, to fill in QL forms and to cooperate fully with the investigator and site personnel
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of orteronel
* Known active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any serious medical illness that could, in the investigator's opinion, potentially interfere with participation in this study
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2014-08-19 (Actual); Study Completion 2034-08-19 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 5 months
  The primary endpoint of the trial is EFS. An event is defined as ONE of the following:
  * death from any cause
  * the presence of radiographic progression AND symptomatic/clinical progression
  * the presence of radiographic progression AND PSA progression
  * the presence of symptomatic/clinical progression AND PSA progression

SECONDARY OUTCOMES:
Adverse events (AEs) | Throughout treatment phase (estimated up to 1 year) until 30 days after last drug administration or prior to start of subsequent anticancer treatment (whichever occurs first)
  All AEs will be assessed according to NCI CTCAE v4.0.
Prostate-specific antigen (PSA) response (30%, 50%, 90% and best) | PSA level at baseline and every 4 weeks until disease progression (estimated up to 1 year)
Time to PSA progression | PSA level at baseline and every 4 weeks until disease progression (estimated up to 1 year)
Radiographic progression-free survival (rPFS) | Every 12 weeks until disease progression (estimated up to 1 year)
Overall survival (OS) | time from trial randomization to the date of death from any cause (estimated up to 4 years)
Quality of Life (QL) | First 6 months of trial treatment
Pain Response | First 6 months of trial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cathomas, MD, Study Chair — Kantonsspital Graubünden; Silke Gillessen, Prof, Study Chair — Cantonal Hospital of St. Gallen
Locations (7):
- Switzerland (7):
  - Kantonsspital Baden, Baden
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Luzern, Luzerne
  - Kantonsspital Muensterlingen, Münsterlingen
  - Kantonsspital - St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun

IPD SHARING:
Plan to Share IPD: No